CLINICAL TRIAL: NCT00867724
Title: A Clinical Study to Evaluate the Performance & Safety of the "Aer-O-Scope" Traveling Through the Colon in Low Risk Subjects
Brief Title: Clinical Study-evaluate Performance&Safety "Aer-O-Scope" in Colon of Low Risk Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GI View Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 190-CLD-AOS
Record Dates: First submitted 2009-03-23; First posted 2009-03-24 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Colon Cancer; Rectal Cancer
Keywords: polyp
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aer-O-Scope Colonoscopy (Experimental): Screening Colonoscopy
  Interventions: Device: Aer-O-Scope Colonoscopy

INTERVENTIONS:
Device: Aer-O-Scope Colonoscopy — Screening Colonoscopy
  Other Names: Aer-O-Scope

SUMMARY:
A double center study to evaluate the safety and efficacy of the Aer-O-Scope in traveling through the colon in low risk subjects.

DETAILED DESCRIPTION:
Asymptomatic adults between the ages of 18 and 70 will undergo screening of the colon using the aer-o-scope, under fluoroscopy, following by screening of the colon using a standard approved colonoscopy for determination of safety.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients between 18 and 70 years of age
* Patients who are generally healthy and classified as low risk for CRC
* Patients who are ready to undergo standard colonoscopy examination including colon prep.
* Signed informed consent

Exclusion Criteria:

* Patients with any known GI related symptoms complaints or GI diseases
* Patients with cancer or other life threatening diseases or conditions
* Patients with unstable or uncontrolled cardiovascular, pulmonary, hepatic, renal' gastrointestinal, genitourinary, hematological, coagulation, immunological, endocrine/metabolic, or other medical disorder that, in the opinion of the investigator, would confound the study results or compromise patient safety. Patients with a known history of blood clotting problems and /or who are on anti-coagulant therapy and cannot stop treatment for the purpose of this study. (Patients taking up to 100mg aspirin for prophylactic treatment are acceptable for this study).
* Pregnant women
* Patients who underwent abdominal surgery that is deemed by the investigator to effect the procedure
* Morbid Obesity (BMI > 40)
* Drug abuse or alcoholism
* Bed-ridden patient
* Inadequate communication with the patient
* Patients under custodial care
* Participation in current clinical study or clinical study within 30 days prior to the procedure

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2009-09; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Ability to screen the entire length of the colon to the cecum. | 30 -60 minutes

SECONDARY OUTCOMES:
Safety endpoints to include incidence of bowel perforation, Colonic bleeding, Damage to colon, rectum and anus mucosa or any other Adverse events | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Erwin M Santo, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No